CLINICAL TRIAL: NCT03259321
Title: Fish, Polyunsaturated Fatty Acids Intake and Type 2 Diabetes in CHNS
Brief Title: Fish, Polyunsaturated Fatty Acids Intake and Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: National Institute of Health and Nutrition (Other Government)
Responsible Party: Principal Investigator, Jingjing Jiao, Associate Professor, Zhejiang University
Other Study IDs: Cohort_PUFA_T2D
Record Dates: First submitted 2017-08-21; First posted 2017-08-23 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Type2 Diabetes
Keywords: Fish; Polyunsaturated fatty acids; CHNS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The role of fishery diet and polyunsaturated fatty acids (PUFA) in the development of type 2 diabetes (T2D) is heavily debated but evidence from large populations in China is scant. The investigators aim to use data from the China Health and Nutrition Survey (CHNS) to assess the long-term association between fish, PUFA intake and T2D risk.

DETAILED DESCRIPTION:
The role of fishery diet and polyunsaturated fatty acids (PUFA) in the development of T2D is heavily debated but evidence from large populations in China is still lacking. The investigators aim to utilize data from China Health and Nutrition Survey (CHNS, 1997-2011). The investigators will calculate cumulative means of fish and PUFA intake based on 3-day food records in each wave. Sex-specific Cox regression models will be used to estimate relative risk of T2D. Results from this work will provide epidemiological evidence for improving recommendations on fish and PUFA intake for Chinese in dietary guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥20 with complete data on diet and follow-up time

Exclusion Criteria:

* Missing information for Type 2 diabetes
* Type 2 diabetes
* Cardiovascular disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CHNS is an ongoing, large-scale, household-based cohort starting in 1989. The survey used a multi-stage, random cluster process to draw a sample of 9 provinces and municipal cities, which take up about half of Chinese population.
Sampling Method: Probability Sample
Enrollment: 15100 (Actual)
Dates: Start 1989-01-01 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Type 2 diabetes | From entry into the study (baseline: 1997-2009) until 2011
  Incidence of type 2 diabetes, on basis of self-reported physician diagnosis, fasting plasma glucose ≥ 7.0 mmol/l or HbA1c ≥ 6.5%

SECONDARY OUTCOMES:
Fish and polyunsaturated fatty acids intake | From entry into the study (baseline: 1997-2009) until 2011
  Cumulative averages of fish and PUFA intake based on 3-day 24-hr recall in each wave

REFERENCES:
- [Derived] Zhuang P, Mao L, Wu F, Wang J, Jiao J, Zhang Y. Cooking Oil Consumption Is Positively Associated with Risk of Type 2 Diabetes in a Chinese Nationwide Cohort Study. J Nutr. 2020 Jul 1;150(7):1799-1807. doi: 10.1093/jn/nxaa103. PMID 32364230
- [Derived] Wu F, Mao L, Zhuang P, Chen X, Jiao J, Zhang Y. Plant-sourced cooking oil consumption is associated with lower total mortality in a longitudinal nationwide cohort study. Clin Nutr. 2020 Dec;39(12):3703-3710. doi: 10.1016/j.clnu.2020.03.031. Epub 2020 Apr 2. PMID 32359931
- [Derived] Zhuang P, Shou Q, Wang W, He L, Wang J, Chen J, Zhang Y, Jiao J. Essential Fatty Acids Linoleic Acid and alpha-Linolenic Acid Sex-Dependently Regulate Glucose Homeostasis in Obesity. Mol Nutr Food Res. 2018 Sep;62(17):e1800448. doi: 10.1002/mnfr.201800448. Epub 2018 Aug 12. PMID 29935107